CLINICAL TRIAL: NCT01719679
Title: Examination of the Effectiveness of Adolescent Vaccines Given in Schools
Brief Title: School Located Adolescent Vaccination Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 08-0204
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-09

CONDITIONS: School Located Vaccine Program
Keywords: school located vaccine program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- School Located Vaccine (SLV) Program (Experimental): A vaccine program carried out by a community vaccinator will be conducted in a limited number of participating schools. The program will be open to the students enrolled at the participating schools
  Interventions: Behavioral: School Located Vaccine (SLV) Program
- no School Located Vaccine (SLV) Program (No Intervention): Schools that are part of the non-intervention arm of the study will not have a school-located vaccine program.

INTERVENTIONS:
Behavioral: School Located Vaccine (SLV) Program — A community vaccinator will administer vaccines to students whose parents consent for their child to participate
  Arms: School Located Vaccine (SLV) Program

SUMMARY:
The provision of adolescent vaccination in a school setting will be feasible and acceptable to parents as evidenced by the number and percentage of students immunized within each school compared to those in schools without a program. The likelihood of vaccination for diphtheria, tetanus, and pertussis (Tdap), human papillomavirus (HPV), and meningococcal conjugate vaccine (MCV4) and all three combined) among eligible students enrolled in schools with a comprehensive school-based immunization program will be significantly higher than that of students enrolled in schools without a school-based immunization program.

ELIGIBILITY:
Inclusion Criteria:

* 2000 (1000 at intervention schools and 1000 in control schools) randomly selected students enrolled in 6th - 8th grade at randomly selected schools
* students who appear to be in need of one or more immunizations of interest at the beginning of the school year
* students enrolled in school by October 1st registration deadline will be included in the analysis

Exclusion Criteria:

* students who appear to have had all immunizations of interest at the beginning of the school year
* students enrolled after the October 1 school registration deadline will be excluded from the analysis
* students enrolled in grades other than 6th, 7th, or 8th grade will not be eligible to participate

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2000 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The likelihood of vaccination among eligible 6th grade students with one or more needed vaccines in intervention schools compared to control schools. | end of the school year 2010 - 2011 compared to beginning of school year 2010 - 2011
  The vaccination status of eligible students enrolled at participating schools will be assessed at the beginning of the school year and at the end of the school year using immunization data from the school, the state registry, community vaccinator registry, and parent records. The assessment will occur in both intervention and control settings.
The likelihood of vaccination among eligible 6th grade students with Tdap vaccine in intervention schools compared to control schools. | end of the school year 2010 - 2011 compared to beginning of school year 2010 - 2011
  The Tdap vaccination status of eligible students enrolled at participating schools will be assessed at the beginning of the school year and at the end of the school year using immunization data from the school, the state registry, community vaccinator registry, and parent records. The assessment will occur in both intervention and control settings.
The likelihood of vaccination among eligible 6th grade students with MCV4 vaccine in intervention schools compared to control schools. | end of the school year 2010 - 2011 compared to beginning of school year 2010 - 2011
  The MCV4 vaccination status of eligible students enrolled at participating schools will be assessed at the beginning of the school year and at the end of the school year using immunization data from the school, the state registry, community vaccinator registry, and parent records. The assessment will occur in both intervention and control settings.
The likelihood of vaccination among eligible 6th grade female students with HPV vaccine in intervention schools compared to control schools. | end of the school year 2010 - 2011 compared to beginning of school year 2010 - 2011
  The HPV vaccination status of eligible female students enrolled at participating schools will be assessed at the beginning of the school year and at the end of the school year using immunization data from the school, the state registry, community vaccinator registry, and parent records. The assessment will occur in both intervention and control settings.

SECONDARY OUTCOMES:
The likelihood of vaccination with Tdap vaccine among eligible 7th and 8th grade students enrolled at intervention schools compared to control schools. | end of the school year 2010 - 2011 compared to beginning of school year 2010 - 2011
  The Tdap vaccination status of students enrolled at participating schools will be assessed at the beginning of the school year and at the end of the school year using immunization data from the school, the state registry, community vaccinator registry, and parent records. The assessment will occur in both intervention and control settings.
The likelihood of vaccination with one or more HPV vaccines among eligible 7th and 8th grade female students enrolled in intervention schools compared to control schools. | end of the school year 2010 - 2011 compared to beginning of school year 2010 - 2011
  The HPV vaccination status of eligible female students enrolled at participating schools will be assessed at the beginning of the school year and at the end of the school year using immunization data from the school, the state registry, community vaccinator registry, and parent records. The assessment will occur in both intervention and control settings.
The likelihood of MCV4 vaccination among eligible 7th and 8th students enrolled in intervention schools compared to control schools. | end of the school year 2010 - 2011 compared to beginning of school year 2010 - 2011
  The MCV4 vaccination status of eligible 7th and 8th grade students enrolled at participating schools will be assessed at the beginning of the school year and at the end of the school year using immunization data from the school, the state registry, community vaccinator registry, and parent records. The assessment will occur in both intervention and control settings.
The likelihood of HPV vaccine series completion among female students in intervention schools compared to control schools. | end of the school year 2010 - 2011 compared to beginning of school year 2010 - 2011
  The HPV vaccine status of female students enrolled at participating schools will be assessed at the beginning of the school year and at the end of the school year using immunization data from the school, the state registry, community vaccinator registry, and parent records. The assessment will occur in both intervention and control settings.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Shlay, MD, MSPH, Principal Investigator — Denver Public Health
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - Kaiser Permanente Colorado, Denver, Colorado